CLINICAL TRIAL: NCT06345287
Title: Response Adaptive Radiotherapy Following Immunotherapy-based Induction for Non-HPV Related Head and Neck Squamous Cell Carcinoma
Brief Title: Response Adaptive Radiotherapy Following Immunotherapy-based Induction for Non-HPV Related HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24/018-4298
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer
Keywords: radical radiotherapy; induction immunotherapy and chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- clinical complete response (Experimental): radiotherapy 60Gy + concurrent chemotherapy + immunotherapy maintenance
  Interventions: Radiation: radical radiotherapy (60Gy); Combination Product: anti-PD-1 or PD-L1 antibody
- deep partial response (Experimental): radiotherapy 66Gy + concurrent chemotherapy + immunotherapy maintenance
  Interventions: Radiation: radical radiotherapy (66Gy); Combination Product: anti-PD-1 or PD-L1 antibody
- non-deep partial response (Experimental): radiotherapy 70Gy+ concurrent chemotherapy + immunotherapy maintenance
  Interventions: Radiation: radical radiotherapy (70Gy); Combination Product: anti-PD-1 or PD-L1 antibody

INTERVENTIONS:
Radiation: radical radiotherapy (60Gy) — concurrent chemoradiotherapy (60Gy) after induction therapy
  Arms: clinical complete response
Radiation: radical radiotherapy (66Gy) — concurrent chemoradiotherapy (66Gy) after induction therapy
  Arms: deep partial response
Radiation: radical radiotherapy (70Gy) — concurrent chemoradiotherapy (70Gy) after induction therapy
  Arms: non-deep partial response
Combination Product: anti-PD-1 or PD-L1 antibody — immunotherapy maintenance with anti-PD-1 or PDL1antibody every three weeks for 1 year after radiotherapy

SUMMARY:
The aim of this study is to develop an adaptive radiation therapy plan for locally advanced head and neck squamous cell carcinoma receiving induction therapy containing immunotherapy and chemotherapy. The therapy plan is based on clinical remission, in order to reduce treatment-related toxic side effects without sacrificing clinical efficacy and improve the quality of life of patients.

DETAILED DESCRIPTION:
Induction chemotherapy combined with immunotherapy has shown promising efficacy in locally advanced head and neck cancers. However, the appropriate dose and range of the following radical radiotherapy treatment remains unknown. Eligibility patients were assigned to three arms depending on the degree of clinical remission: clinical complete response (radiotherapy 60Gy + concurrent chemotherapy + immunotherapy maintenance), deep partial response (radiotherapy 66Gy + concurrent chemotherapy + immunotherapy maintenance, non-deep partial response (radiotherapy 70Gy + concurrent chemotherapy + immunotherapy maintenance). Progression-free survival, overall survival, and treatment-related toxicity would be calculated to evaluate the efficacy of treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Head and neck squamous cell carcinoma patients who undergo 2-4 cycles of induction chemotherapy and immunotherapy and plan to undergo radical radiotherapy treatment ( after MDT evaluation and communication with the patient, surgery is not recommended to preserve organ function, or the patient refuses surgery );
2. Age range from 18 to 75 years old;
3. Squamous cell carcinoma of the head and neck confirmed by pathological tissue biopsy;
4. Clinical staging is T1-2N2-3M0, T3-4N0-3M0 (AJCC 8th edition);
5. HPV or P16 (-);
6. ECOG score 0-1 points;
7. No contraindications to immunotherapy and radiotherapy;
8. The functional level of the main organs meets the following standards:1) The blood routine examination standards need to meet: WBC ≥ 3.0 × 109/L, ANC ≥ 2.0 × 109/L, PLT ≥ 100 × 109/L, HGB ≥ 90g/L (no blood transfusion or blood products within 14 days, no use of G-CSF or other hematopoietic stimulating factors correction);2) Biochemical examination must meet the following standards: TBIL ≤ 2.0 × ULN, ALT, AST ≤ 2.5 × ULN, BUN and CRE ≤ 1.5 × ULN, or endogenous creatinine clearance rate ≥ 60ml/min (Cockcroft Gout formula);3) Good coagulation function: defined as international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; If the subject is receiving anticoagulant treatment, as long as the PT is within the intended range of use of the anticoagulant drug;4) The myocardial enzyme spectrum is within the normal range;
9. Women of childbearing age must have taken reliable contraceptive measures, or have undergone pregnancy tests (serum or urine) within 7 days before enrollment, and the results are negative. They must be willing to use effective methods of contraception during the treatment period and within 2 months thereafter. For male participants whose partners are women of childbearing age, effective methods of contraception should be used during and within 2 months after treatment;
10. Voluntarily participate in this study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Previous or concurrent incurable malignant tumors in other parts, except cured skin basal cell carcinoma, cervical carcinoma in situ, thyroid papillary carcinoma and superficial bladder cancer;
2. Suffering from any active autoimmune disease or having a history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after normal hormone replacement therapy); Asthma patients who suffer from vitiligo or have completely relieved childhood asthma and do not require any intervention in adulthood can be included, while asthma patients who require medical intervention with bronchodilators cannot be included;
3. Suffering from uncontrolled cardiovascular diseases: Grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥ 470 ms); According to NYHA standards, patients with grade III-IV cardiac dysfunction or those with left ventricular ejection fraction (LVEF)<50% indicated by echocardiography; Have experienced myocardial infarction within one year;
4. Active infection or unexplained fever exceeding 38.5 ℃ during screening or before first administration (according to the researcher's judgment, subjects with fever caused by tumors can be included in the study);
5. People with congenital or acquired immune deficiency (such as HIV infected people), active hepatitis B (HBV-DNA ≥ 104 copies/ml) or hepatitis C (hepatitis C antibody is positive, and HCR-RNA is higher than the detection limit of the analytical method);
6. Previously received other PD-1 antibody treatments or other immunotherapies targeting PD-1/PD-L1;
7. Known to be allergic to cisplatin, macromolecular protein preparations, or any anti PD-1 antibody component;
8. If the subject undergoes major surgery without tumor treatment, the toxic reactions and/or complications caused by the surgical intervention must be fully recovered before starting treatment;
9. Pregnant or lactating women;
10. In the investigator's judgment, the subjects had other factors that might have led to their forced discontinuation of the study, such as other serious medical conditions (including mental illness) requiring concomitant treatment, serious abnormalities in laboratory test values, or family or social factors that might have affected the safety of the subjects or the circumstances of the trial data collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first after 2 years of treatment

SECONDARY OUTCOMES:
Overall survival | 2 years
  defined as the time from random assignment to death from any cause or censored at the date of last follow-up
Deep partial response | 2 years
  Defined as maximum tumor diameter retreat ≥ 50%
Local-Regional failure survival | 2 years
  defined as the time from random assignment to documented local or regional relapse, whichever occurred first after 2 years of treatment
Toxicity Adverse events | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) and late radiation toxicities were assessed by NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Junlin Yi, Doctor, Study Chair — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, CAMS & PUMC
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, CAMS & PUMC, Beijing, China